CLINICAL TRIAL: NCT05549622
Title: Impact of a High-Soluble Fiber Diet on the Gut-Muscle Axis in Older Adults
Brief Title: Impact of Diet on the Gut-Muscle Axis in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Jennifer Lee, Principal Investigator, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GRANT13386865
Record Dates: First submitted 2022-08-24; First posted 2022-09-22 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2024-08

CONDITIONS: Sarcopenia; Dietary Exposure; Microbial Colonization
Keywords: skeletal muscle; soluble fiber; gut-muscle axis; microbiome; SCFA; Uremic metabolites
MeSH Terms: conditions — Sarcopenia; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: 24 older adults (> 65y) will be randomized to consume a high- or low-soluble fiber diet
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low-soluble fiber diet (Other)
  Interventions: Other: Low-soluble fiber diet
- High-soluble fiber diet (Active Comparator)
  Interventions: Other: High-soluble fiber diet

INTERVENTIONS:
Other: Low-soluble fiber diet — 12 older adults (>65y) will be randomized to consume the USDA Guidelines for fiber intake (10g of total fiber/1000 calories), as the low-soluble fiber diet
  Arms: Low-soluble fiber diet
Other: High-soluble fiber diet — 12 older adults (>65y) will be randomized to consume 34-35g of total fiber/1000 calories, as the high-soluble fiber diet
  Arms: High-soluble fiber diet

SUMMARY:
Muscle health declines during aging. One factor that may impact muscle health is the community of bacteria that live in our intestines, but studies aimed at improving muscle health by targeting the gut in older adults are sparse. The primary goal of this study is to use a diet that is enriched in soluble fiber, which is exclusively utilized by gut bacteria to make substances that can impact muscle health, to improve muscle-related measures in older adults.

DETAILED DESCRIPTION:
During aging, skeletal muscle mass and physical function decrease, whereas levels of lipids and adipocytes increase within and between muscle cells, thereby worsening muscle composition. As a result of these age-related changes, older adults are at a higher risk for frailty, falls and fracture, disability and hospitalization, and all-cause mortality. Accordingly, elucidation of mechanisms that underlie muscle mass, muscle composition, and physical function, and interventions that positively affect these variables will be important for addressing the public health priority of an improved quality of life and healthy aging in older adults.

The gut microbiome and its metabolic products are involved in mechanisms that impact skeletal muscle mass, muscle composition, and physical function, which has been defined as the gut-muscle axis. For example, muscle mass and physical function are reduced in animals that do not have a microbiome (germ-free mice), and in antibiotic-treated mice, an intervention that reduces gut bacterial content. Investigating further, gut bacteria-derived metabolites affect muscle mass, muscle composition, and physical function in young and aged animals, including positive effects for the short-chain fatty acids (SCFAs) acetate, propionate, and butyrate, and negative effects for indoxyl sulfate (IS) and para-cresol sulfate (PCS). Similarly, phenol sulfate (PS) and phenylacetylglutamine (PAG) are gut microbiome-derived metabolites that were associated with poor muscle composition and worse physical function in studies of older adult humans that were published by our group. Interestingly, higher colonic levels of SCFAs are associated with a lower pH, an important finding because growth of Enterobacteriaceae, a bacterial family that contains genes involved in the production of IS, PCS, PS, and PAG, is limited in an acidic environment and following exposure to physiological levels of SCFAs. Taken together, these data suggest that interventions aimed at increasing bacterial SCFA production may be an important approach for improving muscle-related measures in older adults.

Soluble fiber fermentation by gut bacteria results in the formation of acetate, propionate, and butyrate, and fecal SCFAs proportionally increase, whereas circulating levels of IS and PCS are reduced in response to high-soluble fiber diets. As a proof of concept, fecal and circulating levels of SCFAs, muscle mass, and aerobic exercise capacity were increased in young mice that were fed a relatively higher soluble fiber diet, but few studies have attempted this approach in older adult humans. When considering that fecal levels of SCFAs decrease during aging, whereas plasma levels of IS, PCS, PS, and PAG increase, these data collectively suggest that a high-soluble fiber diet may be an important approach for improving muscle-related measures in older adults humans. To test this hypothesis, older adults will be randomized to consume a high- or low-soluble fiber diet for 12-weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Independently living older adults (> 65y)
2. Sedentary (Godin-Shepard Leisure Time Physical Activity Questionnaire score < 10)
3. Non-smoking
4. Not already consuming a high-fiber diet (> 22, 28 g/day for women, men)
5. Free of gastrointestinal disease (gastrointestinal cancer, inflammatory bowel disease, bariatric surgery, irritable bowel syndrome)
6. Fluent in English
7. Willing to attend three study visits (enrollment, baseline, and week-13)
8. Willing to consume an abundance of fruits, vegetables, nuts/seeds
9. Willing to consume an abundance of soluble fiber-rich foods (broccoli, brussels sprouts, flaxseeds sweetened with dates, lima beans, butternut squash, carrots, collard greens)
10. Willing to tolerate mild gastrointestinal discomfort (bloating, belly grumbling, flatulence). Note that all attempts will be made to replace foods that may trigger these issues.
11. Willing to not consume antibiotics during the 13-week study
12. Willing to not schedule a colonoscopy during the 13-week study

Exclusion Criteria:

1. Unwilling to visit the Tufts Human Nutrition Research Center on Aging (HNRCA) 3x/week to pick up the pre-prepared study diet
2. Unwilling to only consume the provided food (unsweetened tea and/or black coffee are allowed)
3. Food allergies related to foods that are included in the study
4. Chewing problems
5. Unwilling to wear a daily step counter (pedometer)
6. Unwilling to complete a daily questionnaire that will assess gastrointestinal comfort
7. Malnutrition (BMI < 18.5 kg/m2)
8. Use of supplemental probiotics or antibiotics, participation in an investigational drug evaluation, or a recent change in habitual medication use within the 1 month-period prior to the screening visit
9. > 5% weight loss or weight gain within the past 6-months
10. A recent history of alcohol abuse (within the past 5 years)
11. A history of any significant injury or surgery that currently affects physical functioning and ability to perform physical function testing
12. Treatment with immunosuppressive drugs
13. A prior diagnosis of organ failure (heart, liver, renal, respiratory)
14. Diabetes mellitus (type 1, or type 2 with insulin therapy)
15. Chronic kidney disease (eGFR ≤ 30 mL/min/1.73 m2)
16. Overt disease (cancer, dementia, cardiovascular disease)
17. Chronic use of anti-inflammatory medication (corticosteroids)
18. Already enrolled in another research study
19. Active infection, including Tuberculosis , HIV, malaria, hepatitis, shingles, Methicillin-Resistant Staphylococcus Aureus (MRSA), SARS-CoV-2
20. Any major illness or condition that may interfere with study outcomes at the discretion of the study physician
21. Won't remain in Boston for the 13-week study duration
22. Unwilling to complete a daily checklist aimed at quantifying the amount of food eaten on the study diet

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Quantification of SCFAs in fecal samples | Change from baseline when compared with the Week-13 visit
  Fecal levels of bacterial metabolites, including acetate, propionate, and butyrate will be determined at the baseline and week-13 study visits
Quantification of whole-body lean mass with DXA | Change from baseline when compared with the Week-13 visit
  Measurement of whole-body lean mass will be determined at the baseline and week-13 study visits
Quantification of hand grip strength | Change from baseline when compared with the Week-13 visit
  Grip strength will be determined at the baseline and week-13 study visits
Chair stand test | Change from baseline when compared with the Week-13 visit
  The number of chair stands that can be performed in 30 seconds will be determined at the baseline and week-13 study visits

SECONDARY OUTCOMES:
Quantification of thigh muscle composition with computed tomography | Change from baseline when compared with the Week-13 visit
  Determined at the baseline and week-13 study visits
6-minute walk test | Change from baseline when compared with the Week-13 visit
  The distance walked in 6 minutes will be determined at the baseline and week-13 study visits
Quantification of gut bacterial metabolites in plasma | Change from baseline when compared with the Week-13 visit
  Bacterial metabolites, including SCFAs but also indoxyl sulfate, p-cresol sulfate, phenol sulfate, and phenylacetylglutamine will be determined at the baseline and week-13 study visits
Quantification of gut bacterial composition in fecal samples | Change from baseline when compared with the Week-13 visit
  Determined at the baseline and week-13 study visits
Quantification of pH in fecal samples | Change from baseline when compared with the Week-13 visit
  Determined at the baseline and week-13 study visits

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Lustgarten, PhD, Study Director — Scientist II, NEPS Laboratory
Locations (1):
- Jean Mayer Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No data from participants will be shared with researchers not affiliated with this project.